CLINICAL TRIAL: NCT01899638
Title: A Randomized, Open Label, 3 Crossover, Balanced Incomplete Block Study To Evaluate The Pharmacokinetics Of Umeclidinium Bromide and Vilanterol Trifenatate as Monotherapies and Concurrently in Healthy Chinese Subjects.
Brief Title: Pharmacokinetics Of Umeclidinium and Vilanterol in Healthy Chinese, a Randomized, Open Label, 3 Crossover Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115380
Record Dates: First submitted 2013-05-30; First posted 2013-07-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- UMEC/VI 125/25 mcg (Experimental): Combination in high dose
  Interventions: Drug: UMEC/VI 125/25 mcg
- UMEC/VI 62.5/25 mcg (Experimental): Combination in low dose
  Interventions: Drug: UMEC/VI 62.5/25 mcg
- UMEC 125 mcg (Experimental): LAMA mono in high dose
  Interventions: Drug: UMEC 125 mcg
- UMEC 62.5 mcg (Experimental): LAMA mono in low dose
  Interventions: Drug: UMEC 62.5 mcg
- VI 25 mcg (Experimental): LABA mono
  Interventions: Drug: VI 25 mcg

INTERVENTIONS:
Drug: UMEC/VI 125/25 mcg — Combination in high dose
  Arms: UMEC/VI 125/25 mcg
Drug: UMEC/VI 62.5/25 mcg — Combination in low dose
  Arms: UMEC/VI 62.5/25 mcg
Drug: UMEC 125 mcg — LAMA mono in high dose
  Arms: UMEC 125 mcg
Drug: UMEC 62.5 mcg — LAMA mono in low dose
  Arms: UMEC 62.5 mcg
Drug: VI 25 mcg — LABA mono
  Arms: VI 25 mcg

SUMMARY:
This study is to assess the pharmacokinetics (PK), safety and tolerability of UMEC (62.5µg and 125µg) and VI (25µg) as monotherapies and combinations in healthy Chinese subjects.

DETAILED DESCRIPTION:
Vilanterol trifenatate (VI) is a potent and selective long-acting β2 agonist; Umeclidinium bromide (UMEC) is a long-acting, inhaled, muscarinic receptor antagonist (LAMA). Both compounds are in development once daily for the treatment of Chronic Obstructive Pulmonary Disease (COPD).

This study is a randomized, open label, three-period crossover, balanced incomplete block study which will assess the pharmacokinetics (PK), safety and tolerability of UMEC (62.5µg and 125µg) and VI (25µg) as monotherapies and combinations in 20 healthy Chinese subjects. Each subject will receive three of five possible treatments for 10 days each.

Blood samples for PK analysis will be taken at designed timepoints. Safety will be assessed by measurement of ECG QTcF, heart rate, blood pressure, and safety laboratory data and review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females at ratio of 1:1, aged 18 - 45 years . Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Body weight ≥ 50kg and body mass index (weight/height2) within the range of 19 - 24 kg/m2, inclusive.
* Male or female subjects at the time of signing the informed consent:
* Female subject who is child-bearing potential should agree to use one of the contraception methods (contraceptives intrauterine device, implantable progesterone device or oral contraceptive) for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. The subjects must agree to use contraception until completion of the follow-up visit.
* Male subjects have to agree to use one of the contraception methods listed in Section 8.1.2. This criterion is to be followed from the time of the first dose of study medication until completion of the follow-up visit
* Normal systolic (90-139mmHg) and diastolic (60-89mmHg) blood pressure at pre-study screening.
* Subjects who are current non-smokers, who have not used any tobacco products in the 6 month period preceding the screening visit, and have a pack history of 10 pack years. (pack years = (cigarettes per day smoked/20) × number of years smoked)).
* No significant abnormality on 12-lead ECG at screening, QTcF interval must be <450msec (QTcF; machine or manual reading).
* AST (SGOT), ALT (SGPT), and total-bilirubin 1.5xULN at screening. No significant clinical abnormality on other laboratory tests.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subjects who are able to use the inhalation device satisfactorily

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principle investigator or delegate physician deems the subject unsuitable for the study.
* History of mental, cardiac, renal, hepatic, significant gastrointestinal or respiratory disease as judged by the investigator
* A history of breathing problems (i.e. history of asthmatic symptomatology, unless asthma in childhood that has now resolved and no longer requires maintenance therapy which should not be an exclusion).
* A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities. A chest X-ray must be taken at day -1 of the first treatment if a chest X-ray or CT scan is not available within 6 months prior to that day.

History of sensitivity to heparin, heparin-induced thrombocytopenia, or sensitivity to any of the study medications, or components thereof, known allergy or hypersensitivity to milk protein or the excipients lactose monohydrate and magnesium stearate (MgSt), or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

* The subject has taken prescription or non-prescription drugs, including CYP3A/PGP inhibitor, vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Positive result of urine cotinine test.
* The subject has a history of cholecystectomy or biliary tract disease.
* The subject has a significant clinical history or current conditions of glaucoma.
* The subject has a significant clinical history or current conditions of prostatic hypertrophy.
* The subject has a positive pre-study drug screen. A minimum list of drugs that were screened for included amphetamines, barbiturates, cocaine, opiates and benzodiazepines. The detection of drugs with a legitimate medical use was not necessarily an exclusion to study participation. The detection of alcohol was not an exclusion at screening but had to be negative pre-dose and during the study.
* History of regular alcohol consumption within 3 months of the study defined as:
* Abuse of an average weekly intake of greater than 21 units or an average daily intake of greater than three units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than two units (females). One unit was equivalent to a half-pint (220 mL) of beer or one (25 mL) measure of spirits or one glass (125 mL) of wine.
* Female subjects, who are pregnant, planned pregnancy or lactation.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Blood donation or sampled as a study subject within three months preceding the first dose of study drug and blood donation during the entire study in excess of 500mL.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for HIV antibodies.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2013-07-25 (Actual); Study Completion 2013-07-25 (Actual)

PRIMARY OUTCOMES:
Cmax | 5 months
  For both single dose and repeat dose
tmax | 5 months
  For both single dose and repeat dose
tlast | 5 months
  For both single dose and repeat dose
AUC0-t | 5 months
  For both single dose and repeat dose
t1/2 | 5 months
  For both single dose and repeat dose
CL/F | 5 months
  For both single dose and repeat dose
Vd/F | 5 months
  For single dose
AUC0-inf | 5 months
  For single dose
AUC0-t' | 5 months
  For both single dose and repeat dose
C τ | 5 months
  For repeat dose
AUC0-τ | 5 months
  For repeat dose
Ro | 5 months
  For repeat dose
RCmax | 5 months
  For repeat dose
DF | 5 months
  For repeat dose

SECONDARY OUTCOMES:
Blood pressure | 5 months
Heart rate | 5 months
12-lead ECG | 5 months
Chemistry | 5 months
Hematology | 5 months
Urinalysis | 5 months
Adverse event | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hu C, Jia J, Dong K, Luo L, Wu K, Mehta R, Peng J, Ren Y, Gross A, Yu H. Pharmacokinetics and tolerability of inhaled umeclidinium and vilanterol alone and in combination in healthy Chinese subjects: a randomized, open-label, crossover trial. PLoS One. 2015 Mar 27;10(3):e0121264. doi: 10.1371/journal.pone.0121264. eCollection 2015. PMID 25816315
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115380 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115380?search=study&search_terms=115380#rs
- Available data/document: Study Protocol: 115380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115380 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register